CLINICAL TRIAL: NCT07395661
Title: Comparıson Of The Postoperatıve Analgesıc Effıcacy Of Serratus Anterıor Plane Block And Serratus Posterıor Superıor Intercostal Plane Block Performed Under Ultrasonography Guıdance In Vıdeo-Assısted Thoracoscopıc Surgery
Brief Title: Comparison Of Analgesic Methods İn Video-Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Renim Yüksel, Research Assistant, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 225
Record Dates: First submitted 2026-01-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: VATS; Pain Management; Plane Blocks
Keywords: VATS; Pain Management; Plane Blocks; SPSIPB; SAPB
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SERRATUS ANTERİOR PLANE BLOCK (Experimental): Patients in this group received an ultrasound-guided serratus anterior plane block for postoperative analgesia following video-assisted thoracoscopic surgery.
  Interventions: Procedure: Ultrasound guided serratus anterior plane block
- SERRATUS POSTERİOR SUPERİOR İNTERCOSTAL PLANE BLOCK (Experimental): Patients in this group received an ultrasound-guided serratus posterior superior intercostal plane block for postoperative analgesia following video-assisted thoracoscopic surgery.
  Interventions: Procedure: Ultrasound guided serratus posterior superior intercostal plane block

INTERVENTIONS:
Procedure: Ultrasound guided serratus anterior plane block — An ultrasound-guided serratus anterior plane block was performed for postoperative analgesia in patients undergoing video-assisted thoracoscopic surgery.
  Arms: SERRATUS ANTERİOR PLANE BLOCK
Procedure: Ultrasound guided serratus posterior superior intercostal plane block — An ultrasound-guided serratus posterior superior intercostal plane block was performed for postoperative analgesia in patients undergoing video-assisted thoracoscopic surgery.
  Other Names: Serratus posterior superior intercostal plane block
  Arms: SERRATUS POSTERİOR SUPERİOR İNTERCOSTAL PLANE BLOCK

SUMMARY:
Comparison of the Analgesic Efficacy of Serratus Anterior Plane Block and Serratus Posterior Superior Intercostal Plane Block in Patients Undergoing Video-Assisted Thoracoscopic Surgery Introduction and Objective: The aim of this study is to compare the postoperative analgesic efficacy of the serratus anterior plane block and serratus posterior superior intercostal plane block performed under ultrasonography guidance in patients undergoing video-assisted thoracoscopic surgery.

Patients with ASA grades I-III, aged 18-65, will be included in the study. Standard general anesthesia will be administered to the patients. Postoperative analgesia evaluation will be conducted using VAS and NRS scores at specific time points after surgery Additional analgesic requirements and patient satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 65 years ASA physical status I-III Scheduled for elective video-assisted thoracoscopic surgery (VATS) Provided written information consent

Exclusion Criteria:

* History of allergy or toxicity to local anesthetic agents
* Known or suspected coagulopathy
* Infection at the site of block injection
* Advanced organ failure
* Diagnosed mental retardation
* Pregnancy
* Pediatric patients
* History of thoracotomy
* Requirement for postoperative intubation
* Emergency surgery
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | At postoperative 30 minute and 1, 4, 8, 12, 24 hours
  Postoperative pain intensity was assessed using the Visual Analog Scale (VAS) where 0 indicates no pain and 10 indicates the worst imaginable pain

SECONDARY OUTCOMES:
Postoperative pain intensity assessed by Numeric Rating Scale (NRS) | 30 minutes, 1, 4, 8, 12, 24 hours after surgery
  Postoperative pain intensity will be assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Siences Gazi Yasargil Training and Research Hospital, Diyarbakır, Kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No